CLINICAL TRIAL: NCT04857112
Title: A Phase 2, Randomized, Double-Blinded, Placebo Controlled, Parallel Group Study Evaluating the Efficacy and Safety of Amiselimod (MT-1303) in Subjects With Mild to Moderate Ulcerative Colitis (UC)
Brief Title: Study Evaluating Efficacy and Safety of Amiselimod (MT-1303) in Mild to Moderate Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMUC-2023
Record Dates: First submitted 2021-04-19; First posted 2021-04-23 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — amiselimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose (Experimental): MT-1303 loading dose of 0.4 mg once daily (QD) (Day 1-14) then maintenance dose of 0.2 mg QD (Day 15-85)
  Interventions: Drug: Low Dose MT-1303
- High Dose (Experimental): MT-1303 loading dose of 0.8 mg QD (Day 1-14) then maintenance dose of 0.4 mg QD (Day 15-85)
  Interventions: Drug: High Dose MT-1303
- Placebo (Placebo Comparator): Matching placebo, QD (Day 1-85)
  Interventions: Drug: Placebo
- Open Label Extension Period (Other): 0.4 mg MT-1303 QD for 36 weeks for those participants who continue on to the OLE period from the double-blind portion of the clinical study
  Interventions: Drug: MT-1303

INTERVENTIONS:
Drug: Low Dose MT-1303 — MT-1303 loading dose of 0.4 mg once daily (QD) (Day 1-14) then maintenance dose of 0.2 mg QD (Day 15-85)
  Other Names: Amiselimod
  Arms: Low Dose
Drug: High Dose MT-1303 — MT-1303 loading dose of 0.8 mg QD (Day 1-14) then maintenance dose of 0.4 mg QD (Day 15-85)
  Other Names: Amiselimod
  Arms: High Dose
Drug: Placebo — Matching placebo, QD (Day 1-85)
  Other Names: Amiselimod
  Arms: Placebo
Drug: MT-1303 — 0.4 mg MT-1303 QD for 36 weeks for those participants who continue on to the OLE period from the double-blind portion of the clinical study
  Other Names: Amiselimod
  Arms: Open Label Extension Period

SUMMARY:
The study will assess the efficacy and safety of oral MT-1303 compared to placebo at 12 weeks as the induction treatment in subjects with active mild to moderate ulcerative colitis (UC), as well as maintenance treatment with open-label MT-1303 for up to 36 weeks.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blinded, placebo-controlled 3-arm, multi-center, parallel-group study with an open-label extension (OLE) period. The study includes a Screening Period (of up to 28 days) and a 12-week Double-Blind Period (Day 1 through Day 85) for all subjects. Subjects completing the Double-Blind Period through Day 85 will be provided the opportunity to continue in the OLE Period of the study to receive treatment through approximately one year. Subjects who do not participate in the OLE Period will be followed for 84 days in a Safety Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if they are male or female aged between 18 to 75 years at time of consent (inclusive) with normal vital signs and a diagnosis of active mild ulcerative colitis (UC) (modified Mayo Score of 3 or 4) or moderate UC (modified Mayo Score of 5 to 8) confirmed at least 12 weeks prior to randomization by clinical and endoscopic evidence and corroborated by a histopathology report.
* Subjects must have an endoscopic subscore of ≥2 from and evidence of active UC extending ≥15 cm from the anal verge confirmed by a screening colonoscopy.
* If subjects are receiving oral or rectal 5-aminosalicylates (5-ASAs) or oral corticosteroids (≤20 mg prednisolone equivalent) for treatment of their UC, they must be on a stable dose for at least 28 days prior to randomization.
* Subjects who complete the Double-Blind Period of the study who, in the opinion of the Investigator, would benefit from continued treatment, may participate in the Open Label Extension (OLE) Period.

Exclusion Criteria:

* Any of the following: a diagnosis of Crohn's disease, indeterminate colitis, colitis (pseudomembranous, microscopic, or ischemic) or coeliac disease, current or recent (within 12 weeks prior to randomization) evidence of fulminant colitis, proctitis (defined as a rectal inflammation within 15 cm from the anal verge), abdominal abscess, toxic megacolon, bowel obstruction, or bowel perforation; a history or evidence of any colonic resection or subtotal or total colectomy, ileostomy, colostomy, known fixed symptomatic stenosis of the intestine, unresected adenomatous colonic polyps, or colonic mucosal dysplasia.
* Clinically significant infections (e.g., pneumonia, pyelonephritis, or septicemia) within 4 weeks prior to randomization or previous clinically significant infections requiring hospitalization within 6 months prior to randomization, active or latent tuberculosis, infections of hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or previous shingles outbreak.
* Active SARS-CoV-2 infection or complications related to COVID-19.
* A history of, or currently active, primary or secondary immunodeficiency, presence of progressive multifocal leukoencephalopathy (PML), or presence of demyelinating diseases.
* A history or evidence of two or more failures with biologic treatment for UC.
* Currently taking any medication for treatment of UC other than oral or rectal 5-ASAs (5-aminosalicylic acids) or oral corticosteroids (≤20 mg prednisolone equivalent)
* Been taking enemas or suppositories (other than stable dose of 5-ASA) for treatment of UC within 2 weeks prior to the Screening Visit.
* Been taking an unstable dose of probiotics or antidiarrheals 2 weeks prior to the Screening Visit.
* Had recent myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure with hospitalization, Class III/IV heart failure, Mobitz Type II 2nd degree or 3rd degree atrioventricular (AV) block, sick sinus syndrome, prolonged QT interval, Wolff Parkinson White or other conduction abnormalities, low heart rate, ongoing treatment with Class I or Class III anti-arrhythmic drugs, heart-rate-lowering calcium-channel blockers, β blockers or with any other drugs which can reduce the heart rate, have known high risk for QT/QTc prolongation, or have clinically significant abnormal findings in 12-lead ECG that the Investigator considers may jeopardize the subject's health.
* Forced expiratory volume in one second (FEV1) or forced expiratory vital capacity (FVC) <70% of predicted values at screening. For sites where DLCO (diffusing capacity of the lungs for carbon monoxide) will be assessed, the value (mL/min/mmHg) is < 80% of the predicted normal value for age, height, and gender.
* Macular oedema as assessed by OCT (Optical Coherence Tomography).
* History of non-response or treatment failure with MT-1303 or other sphingosine 1 phosphate (S1P) receptor modulators.
* Fecal microbiota transplantation (FMT) within 12 months prior to the Screening Visit.
* Any of the following laboratory abnormalities:

  * Hemoglobin (Hb) <9.0 g/dL.
  * White blood cell (WBC) count <3.50 × 109/L (<3,500/µL).
  * Neutrophil count <1.50 × 109/L (<1,500/µL).
  * Lymphocyte count <0.80 × 109/L (<800/µL).
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >2 × the upper limit of normal (ULN).
  * Bilirubin >1.5 x the ULN; subjects with Gilbert's syndrome may be enrolled with total bilirubin up to 5.0 mg/dl.
* Positive stool tests for enteric pathogens, pathogenic ova or parasites, or Clostridium difficile (C. difficile) during the Screening Period. If subject has a history of recent C. difficile infection (within 60 days prior to Screening Visit), they should not be considered for study enrollment until subject has been treated for C. difficile and is symptom free for at least 14 days prior to the Screening Visit.
* Any physical or mental conditions which would interfere with the study participation, collection of data, or study completion as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-11-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the modified Mayo Score at Day 85 | Baseline to Day 85
  The modified Mayo Score for ulcerative colitis disease activity provides an assessment of disease severity and can be used to monitor subjects during therapy. Scoring is accomplished by summation of subscores for endoscopic findings, stool frequency, and rectal bleeding, with higher scores indicating worse severity. Each subscore ranges from 0 to 3. The modified Mayo Score is defined as the sum of the endoscopy findings subscore + stool frequency subscore + rectal bleeding subscore, with a range from 0 to 9.

SECONDARY OUTCOMES:
The proportion of subjects with endoscopic improvement at Day 85 | Baseline to Day 85
  The Mayo endoscopic subscore ranges from 0 to 3, with higher scores indicating worse severity. Endoscopic improvement is a Mayo endoscopic subscore of ≤1.
The change from Baseline in the 2-component Mayo Score at Day 85. | Baseline to Day 85
  2-component Mayo scoring is accomplished by summation of subscores for endoscopic findings and rectal bleeding, with higher scores indicating worse severity. Each subscore ranges from 0 to 3. The 2-component Mayo Score is the sum of the rectal bleeding plus endoscopic subscores, with a range from 0 to 6.
The proportion of subjects with clinical remission at Day 85 based on the modified Mayo Score | Baseline to Day 85
  The modified Mayo Score for ulcerative colitis disease activity provides an assessment of disease severity and can be used to monitor subjects during therapy. Scoring is accomplished by summation of subscores for endoscopic findings, stool frequency, and rectal bleeding, with higher scores indicating worse severity. Each subscore ranges from 0 to 3.
  Remission is defined as follows:
  * Endoscopy subscore of ≤1 (excludes friability); and
  * Rectal bleeding subscore of 0; and
  * At least one-point decrease in stool frequency subscore from Baseline to achieve a stool frequency subscore of ≤1.

CONTACTS AND LOCATIONS:
Overall Officials: John Lahey, Study Director — Bausch Health Americas, Inc.
Locations (185):
- United States (22):
  - Bausch Site 025, Chandler, Arizona
  - Salix Site 004, Los Angeles, California
  - Salix Site 003, Rancho Cucamonga, California
  - Salix Site 007, Rialto, California
  - Salix Site 006, Ventura, California
  - Bausch Site 013, Maitland, Florida
  - Bausch Site 024, Miami, Florida
  - Salix Site 005, Miramar, Florida
  - Bausch site 026, Orlando, Florida
  - Salix Site 010, Snellville, Georgia
  - Bausch Site 011, Chicago, Illinois
  - Bausch Site 020, Glenview, Illinois
  - Bausch Site 008, Lafayette, Louisiana
  - Bausch Site 022, Metairie, Louisiana
  - Salix Site 001, Shreveport, Louisiana
  - Salix Site 002, Freehold, New Jersey
  - Bausch Site 017, Mentor, Ohio
  - Bausch Site 021, Oklahoma City, Oklahoma
  - Bausch Site 014, El Paso, Texas
  - Bausch Site 018, Houston, Texas
  - Bausch Site 019, Houston, Texas
  - Bausch Site 012, Suffolk, Virginia
- Australia (5):
  - Bausch site 1005, Adelaide
  - Bausch site 1001, Brisbane
  - Bausch site 1006, Epping
  - Bausch site 1002, South Brisbane
  - Bausch site 1007, Woolloongabba
- Belarus (4):
  - Bausch Site 1101, Homyel
  - Bausch Site 1104, Minsk
  - Bausch Site 1103, Mogilev
  - Bausch Site 1105, Vitebsk
- Bulgaria (7):
  - Bausch Site 1301, Sofia
  - Bausch Site 1304, Sofia
  - Bausch Site 1302, Sofia
  - Bausch Site 1307, Sofia
  - Bausch Site 1303, Sofia
  - Bausch Site 1305, Stara Zagora
  - Bausch Site 1306, Varna
- Czechia (6):
  - Bausch Health Site 1404, Brno
  - Bausch Health Site 1405, Hradec Králové
  - Bausch Health Site 1403, Olomouc
  - Bausch Health Site 1406, Pardubice
  - Bausch Health Site 1401, Prague
  - Bausch Health Site 1402, Slaný
- Estonia (3):
  - Bausch Site 1503, Pärnu
  - Bausch Site 1501, Tallinn
  - Bausch Site 1502, Tallinn
- Georgia (6):
  - Bausch Health Site 1602, Tbilisi
  - Bausch Health Site 1603, Tbilisi
  - Bausch Health Site 1604, Tbilisi
  - Bausch Health Site 1605, Tbilisi
  - Bausch Health Site 1606, Tbilisi
  - Bausch Health Site 1601, Tbilisi
- Germany (15):
  - Bausch Health Site 1718, Augsburg
  - Bausch Health Site 1705, Berlin
  - Bausch Health Site 1716, Berlin
  - Bausch Health Site 1717, Brandenburg
  - Bausch Health Site 1708, Cologne
  - Bausch Health Site 1710, Dresden
  - Bausch Health Site 1707, Frankfurt am Main
  - Bausch Health Site 1706, Kiel
  - Bausch Health Site 1712, Mainz
  - Bausch Health Site 1713, Mannheim
  - Bausch Health Site 1702, Nordhausen
  - Bausch Health Site 1709, Remscheid
  - Bausch Health Site 1714, Rostock
  - Bausch Health Site 1701, Tübingen
  - Bausch Health Site 1703, Wipperfürth
- Hungary (4):
  - Bausch Health Site 1805, Békéscsaba
  - Bausch Health Site 1803, Kistarcsa
  - Bausch Health Site 1801, Mohács
  - Bausch Health Site 1802, Székesfehérvár
- Italy (7):
  - Bausch Health Site 1906, Florence
  - Bausch Health Site 1904, Messina
  - Bausch Health Site 1909, Milan
  - Bausch Health Site 1901, Milan
  - Bausch Health Site 1908, Monza
  - Bausch Health Site 1907, Padua
  - Bausch Health Site 1903, Turin
- Japan (21):
  - Bausch Health Site 2004, Chiba
  - Bausch Health Site 2014, Chiba
  - Bausch Health Site 2011, Fukuoka
  - Bausch Health Site 2005, Hiroshima
  - Bausch Health Site 2009, Hokkaido
  - Bausch Health Site 2019, Hokkaido
  - Bausch Health Site 2016, Hyōgo
  - Bausch Health Site 2013, Iwata
  - Bausch Health Site 2020, Kagawa
  - Bausch Health Site 2022, Kamakura
  - Bausch Health Site 2017, Mie
  - Bausch Health Site 2002, Miyagi
  - Bausch Health Site 2008, Nagasaki
  - Bausch Health Site 2006, Ōita
  - Bausch Health Site 2007, Saga
  - Bausch Health Site 2023, Takayama
  - Bausch Health Site 2012, Tokyo
  - Bausch Health Site 2018, Tokyo
  - Bausch Health Site 2010, Tokyo
  - Bausch Health Site 2021, Tokyo
  - Bausch Health Site 2003, Tokyo
- Moldova (5):
  - Bausch Health Site 2202, Chisinau
  - Bausch Health Site 2205, Chisinau
  - Bausch Health Site 2201, Chisinau
  - Bausch Health Site 2203, Chisinau
  - Bausch Health Site 2204, Chisinau
- Poland (22):
  - Bausch Health Site 2320, Bialystok
  - Bausch Health Site 2309, Bydgoszcz
  - Bausch Health Site 2323, Elblag
  - Bausch Health Site 2301, Krakow
  - Bausch Health Site 2306, Krakow
  - Bausch Health Site 2314, Lodz
  - Bausch Health Site 2318, Nowy Targ
  - Bausch Health Site 2305, Oświęcim
  - Bausch Health Site 2316, Rzeszów
  - Bausch Health Site 2304, Sopot
  - Bausch Health Site 2321, Staszów
  - Bausch Health Site 2302, Szczecin
  - Bausch Health Site 2315, Tychy
  - Bausch Health Site 2311, Warsaw
  - Bausch Health Site 2303, Warsaw
  - Bausch Health Site 2322, Warsaw
  - Bausch Health Site 2308, Warsaw
  - Bausch Health Site 2310, Wierzchosławice
  - Bausch Health Site 2313, Wroclaw
  - Bausch Health Site 2317, Wroclaw
  - Bausch Health Site 2307, Wroclaw
  - Bausch Health Site 2319, Wroclaw
- Russia (17):
  - Bausch Health Site 2403, Barnaul
  - Bausch Health Site 2416, Chelyabinsk
  - Bausch Health Site 2417, Chita
  - Bausch Health Site 2419, Moscow
  - Bausch Health Site 2406, Moscow
  - Bausch Health Site 2405, Nizhny Novgorod
  - Bausch Health Site 2411, Novosibirsk
  - Bausch Health Site 2421, Orenburg
  - Bausch Health Site 2413, Pyatigorsk
  - Bausch Health Site 2408, Saint Petersburg
  - Bausch Health Site 2409, Saint Petersburg
  - Bausch Health Site 2415, Saint Petersburg
  - Bausch Health Site 2402, Saint Petersburg
  - Bausch Health Site 2422, Samara
  - Bausch Health Site 2410, Tomsk
  - Bausch Health Site 2401, Veliky Novgorod
  - Bausch Health Site 2423, Yekaterinburg
- Serbia (5):
  - Bausch Health Site 2501, Belgrade
  - Bausch Health Site 2502, Belgrade
  - Bausch Health Site 2503, Belgrade
  - Bausch Health Site 2505, Kragujevac
  - Bausch Health Site 2504, Pančevo
- Slovakia (6):
  - Bausch Health Site 2601, Banská Bystrica
  - Bausch Health Site 2604, Bratislava
  - Bausch Health Site 2605, Brezno
  - Bausch Health Site 2603, Košice
  - Bausch Health Site 2602, Prešov
  - Bausch Health Site 2606, Rimavská Sobota
- South Korea (12):
  - Bausch Health Site 2109, Busan
  - Bausch Health Site 2112, Daegu
  - Bausch Health Site 2105, Daegu
  - Bausch Health Site 2114, Daegu
  - Bausch Health Site 2107, Seoul
  - Bausch Health Site 2101, Seoul
  - Bausch Health Site 2110, Seoul
  - Bausch Health Site 2102, Seoul
  - Bausch Health Site 2103, Seoul
  - Bausch Health Site 2108, Seoul
  - Bausch Health Site 2113, Suwon
  - Bausch Health Site 2106, Wŏnju
- Taiwan (4):
  - Bausch Health Site 2703, Kaohsiung City
  - Bausch Health Site 2702, Taichung
  - Bausch Health Site 2701, Taichung
  - Bausch Health Site 2704, Tainan
- Ukraine (14):
  - Bausch Health Site 2815, Ivano-Frankivsk
  - Bausch Health Site 2803, Kharkiv
  - Bausch Health Site 2801, Khmelnytskyi
  - Bausch Health Site 2804, Kyiv
  - Bausch Health Site 2807, Kyiv
  - Bausch Health Site 2806, Kyiv
  - Bausch Health Site 2814, Kyiv
  - Bausch Health Site 2811, Lutsk
  - Bausch Health Site 2810, Lviv
  - Bausch Health Site 2805, Odesa
  - Bausch Health Site 2816, Vinnytsia
  - Bausch Health Site 2812, Zaporizhia
  - Bausch Health Site 2808, Zaporizhia
  - Bausch Health Site 2802, Zhytomyr

IPD SHARING:
Plan to Share IPD: Undecided